CLINICAL TRIAL: NCT00589862
Title: Clinical Management of Antiplatelet Drug Resistance in Patients With Drug Eluting Coronary Stents
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to secure adequate funding
Sponsor: Creighton University (Other)
Responsible Party: Daniel Hilleman, PharmD, Creighton University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-14622; 07-14622
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stents; Clopidogrel Resistance; Aspirin Resistance
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Plavix (Clopidogrel)

INTERVENTIONS:
Drug: Plavix (Clopidogrel) — 150 mg tablet of Plavix (Clopidogrel) per day for 12 months if resistance is identified

SUMMARY:
It is recommended that patients who have drug-eluting stents placed in their coronary arteries take aspirin and Plavix (Clopidogrel) for at least a year. Patients who stop taking these antiplatelet drugs or who have resistance to the antiplatelet effects of these drugs are at a higher risk of clots occurring inside the stents which may result in a heart attack. At the present time, it is unknown if increasing the doses of the antiplatelet agents is effective in overcoming this resistance. The purpose of this project is to identify patients with antiplatelet drug resistance and to test whether an increase in the Plavix (Clopidogrel) dose overcomes antiplatelet drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Required Coronary Artery Angioplasty with a drug-eluting stent deployment

Exclusion Criteria:

* The last drug-eluting stent placed greater than 2 weeks prior
* Aspirin or Plavix (Clopidogrel) allergy or contraindication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
to evaluate the frequency of aspirin and Plavix (Clopidogrel) resistance (as measured by a percent inhibition of platelet aggregation) in patients undergoing coronary drug-eluting stent deployment | 3 month intervals up to 12 months

SECONDARY OUTCOMES:
to assess if a Plavix (Clopidogrel) dose increase in patients with resistance to both aspirin and Plavix (Clopidogrel) is effective in overcoming antiplatelet drug resistance | 3 month intervals up to 12 months
to evaluate the frequency of major adverse cardiovascular events in patients with and without antiplatelet resistance and following a dose increase in Plavix (Clopidogrel). | 3 month intervals up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hilleman, PharmD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States